CLINICAL TRIAL: NCT04166214
Title: Oral Pathology Asynchronous Telementoring Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-01268
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dental Providers (Experimental): The tele-mentoring intervention involves training dental faculty members and residents to use intraoral cameras to take photographs of oral lesions and place them in the Dentrix electronic health record (EHR), along with descriptions of the lesions.
  Interventions: Other: Imaging using intraoral cameras
- Dental Patients (Experimental): The tele-mentoring intervention involves training dental faculty members and residents to use intraoral cameras to take photographs of oral lesions and place them in the Dentrix electronic health record (EHR), along with descriptions of the lesions.
  Interventions: Other: Imaging using intraoral cameras

INTERVENTIONS:
Other: Imaging using intraoral cameras — The SOPROCARE is intended for clinical practice of general dentistry, as an aid in the diagnosis of pit and fissure caries, as an aid to highlight dental plaque and gingival inflammations and as intra-oral camera to visualize anatomical details that are invisible to the naked eye or with a mirror. In CARIO mode, the camera helps the dental practitioner to highlight carious warning on pits and fissures of the occlusal side of the teeth. In DAYLIGHT mode, the camera enables you to visualize anatomical details invisible to the naked eye or with a mirror. In PERIO mode, the camera helps the dental practitioner to see the presence of dental plaque but also to highlight gingival inflammations . This mode offers to the dentist and/or hygienist a tool for an improved communication, motivation and education of his/her patients, who will then become aware of their oral health condition.
  Other Names: Aceton Soprocare Intraoral Camera

SUMMARY:
The purpose of the proposed research project is to evaluate and enhance the feasibility and acceptability of integrating a tele-mentoring component into the identification of oral lesions at the 6 dental clinics of Family Health Centers at NYU Langone (FHC), a Federally Qualified Health Center (FQHC) in Brooklyn, NY.

DETAILED DESCRIPTION:
The tele-mentoring intervention involves training dental faculty members and residents to use intraoral cameras to take photographs of oral lesions and place them in the Dentrix electronic health record (EHR), along with descriptions of the lesions. Using a mixed-methods approach, the study will evaluate and enhance the feasibility and acceptability of integrating a tele-mentoring component into the identification of oral lesions at the 6 FHC dental clinics.

ELIGIBILITY:
Inclusion Criteria:

Dental patients will be eligible for study participation if they meet the following criteria:

1. Greater than or equal to 18 years of age.
2. Live in any of the 5 boroughs of New York, NY and visit a participating FHC dental clinic for routine dental care.
3. Able and willing to provide informed consent, have their oral lesion(s) photograph(s) and accompanying data entered into the Dentrix EHR, and participate in an exit interview.

Dental providers will be eligible for study participation if they meet the following criteria:

1. Greater than or equal to 18 years of age.
2. Be employed as a dentist or placed as a dental resident at a participating FHC dental clinic.
3. Able and willing to provide informed consent and participate in feasibility testing (provider survey or semi-structured interview).

Exclusion Criteria:

Dental patients will be excluded from study participation if they meet the following criteria:

1. Have an acute or terminal illness or a serious mental illness or any other severe health condition(s) that might preclude visiting an oral health care provider.
2. Are currently participating in another oral health study.

Dental providers will be excluded from study participation if they meet the following criteria:

1. Have an acute or terminal illness or a serious mental illness or any other severe health condition(s) that might preclude them from completing the feasibility testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Mohadjeri-Franck, DMD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health Dental Medicine, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Access Criteria: The investigator who proposed to use the data. Requests should be directed to Natalie.Mohadjeri-Franck@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dental Providers | Dental Patients
Started | 12 | 39
Completed | 12 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dental Providers | Dental Patients | Total
Number analyzed (Participants) | 12 | 39 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (1.4) | 40.9 (20.6) | 37.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 2 | 19 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 25 | 26
  Not Hispanic or Latino | 11 | 7 | 18
  Unknown or Not Reported | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 32 | 33
Region of Enrollment [Number; unit: participants]
  United States | 12 | 39 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Dental Patients Who Strongly Agreed or Agreed That the Use of an Intra-Oral Camera By Their Dentists Helped Them to Better Understand Oral Cancer Screening
Description: Consented patients will be asked to complete a brief Patient Exit Survey (5 statements) at the end of their dental appointments after being screened for oral cancer lesions using an intraoral camera. Responses to the second statement are reported for this outcome measure. The statement is scored on a Likert Scale from 1 - Strongly Disagree to 5 - Strongly Agree.
Time Frame: At the end of the dental appointment, 30-45 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Dental Patients
Number analyzed (Participants) | 39
percentage of participants | 94.9

2. Primary Outcome: Percentage of Dental Patients Who Strongly Agreed or Agreed That Dentists Answered Their Questions About Oral Cancer and Were Able to Provide Them With Resources
Description: Consented patients will be asked to complete a brief Patient Exit Survey (5 statements) at the end of their dental appointments after being screened for oral cancer lesions using an intraoral camera. Responses to the fourth statement are reported for this outcome measure. The statement is scored on a Likert Scale from 1 - Strongly Disagree to 5 - Strongly Agree.
Time Frame: At the end of the dental appointment, 30-45 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Dental Patients
Number analyzed (Participants) | 39
percentage of participants | 94.8

3. Secondary Outcome: Percentage of Dental Providers Who Reported Successfully Providing the Tele-Mentoring Intervention
Description: Dentists are given a Provider "Essential Components" Checklist to fill out. This checklist summarizes the essential components of incorporating a tele-mentoring intervention into the identification of oral lesions via use of intraoral cameras to take photographs of oral lesions at chairside, uploading them into Dentrix, and conferring with an oral pathology expert.
  Successful provision of the intervention is indicated by marking "item met" for all 10 intervention elements listed in the checklist.
Time Frame: At the end of the dental appointment, 30-45 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Dental Providers
Number analyzed (Participants) | 12
percentage of participants | 100

4. Secondary Outcome: Percentage of Dental Providers Who Reported That The Process Was Clear and Straightforward
Description: The process includes from EHR data entry to interaction with the oral surgeon over findings to patient referral
Time Frame: At the end of the dental appointment, 30-45 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Dental Providers
Number analyzed (Participants) | 12
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: At the end of the dental appointment, 30-45 minutes
Arm/Group | Dental Providers | Dental Patients
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/39
Other Adverse Events (participants affected / at risk) | 0/12 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT04166214/Prot_SAP_000.pdf